CLINICAL TRIAL: NCT00511264
Title: Prospective Evaluation of the Impact of Laparoscopic Ultrasound (LUS) Guided Fine-Needle Aspiration or Tru-Cut Biopsy in Patients With Upper GI Tract Cancer
Brief Title: Laparoscopic Ultrasound Guided Tissue Sampling in Patients With Cancer of the Upper Gastrointestinal Tract
Status: Completed | Type: Observational
Sponsor: Odense University Hospital (Other)
Other Study IDs: 2007-10
Record Dates: First submitted 2007-08-01; First posted 2007-08-03 (Estimated); Last update posted 2008-05-29 (Estimated); Status verified 2008-05

CONDITIONS: Esophageal Cancer; Gastric Cancer; Pancreatic Cancer; Liver Cancer
Keywords: Laparoscopy; Ultrasound; Cancer; Biopsy
MeSH Terms: conditions — Esophageal Neoplasms; Stomach Neoplasms; Pancreatic Neoplasms; Liver Neoplasms; Neoplasms

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Laparoscopic Ultrasound (LUS) is an important part of the pre-treatment evaluation of patients with upper gastrointestinal tract cancer (esophageal, gastric, pancreatic and liver cancer). When a suspect lesion is visualized during LUS a biopsy should be provided in order to differentiate between benign and malignant lesions. A new system for LUS guided biopsy has been developed, but how often these biopsies are clinically relevant (i.e. changing patient management)and how reliable are these biopsies are unknown.

The study hypothesis is that LUS guided biopsies are accurate and clinically relevant in the pre-treatment evaluation of patients with upper gastrointestinal tract cancer.

ELIGIBILITY:
Inclusion Criteria:

* Biopsy proven upper GI tract cancer
* Laparoscopic Ultrasound indicated during pre-treatment evaluation

Exclusion Criteria:

* Patients unfit for surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2007-05; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael B Mortensen, MD, Ph.D., Principal Investigator — Department of Surgery, Odense University Hospital
Locations (1):
- Department of Surgery, Odense University Hospital, Odense, Denmark